CLINICAL TRIAL: NCT02682901
Title: Impact of Timed Bromocriptine-QR Therapy Upon Measures of Sympathetic Tone and Vascular Biology in Type 2 Diabetes Subjects
Brief Title: Bromocriptine-QR Therapy on Sympathetic Tone and Vascular Biology in Type 2 Diabetes Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Principal Investigator, Elias S Siraj, Professor of Medicine Chief, Division of Endocrine and Metabolic Disorders Director, Strelitz Diabetes Center Associate Dean for Clinical Research, Eastern Virginia Medical School
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-06-FB-0119
Record Dates: First submitted 2016-02-04; First posted 2016-02-17 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Autonomic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Bromocriptine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cycloset (Bromocriptine-QR) (Active Comparator): Subjects will be randomized in a 1:1 ratio to receive UDT (usual diabetes therapy) plus bromocriptine-QR. Following randomization subjects will be titrated to the maximum tolerated dose of the study drug over a four-week period. During these first 4 weeks, the daily dose of the study drug will be titrated up by one tablet (0.8 mg bromocriptine-QR) per day on a weekly basis until a maximal tolerated dose of at least two tablets (1.6 mg/day bromocriptine-QR) and no more than four tablets (3.2 mg/per day b-QR) is achieved. Subjects will be maintained at their maximum tolerated dose of between two to four tablets per day (1.6 to 3.2 mg bromocriptine-QR per day) for the duration of the study. Subjects will be seen at 4 weeks after randomization, at 12 weeks after randomization, and then at study end (week 24 or early termination).
  Interventions: Drug: Cycloset
- Placebo (Placebo Comparator): Subjects will be randomized in a 1:1 ratio to receive UDT (usual diabetes therapy) plus placebo. Following randomization subjects will be titrated to the maximum tolerated dose of the study drug over a four-week period. During these first 4 weeks, the daily dose of the study drug will be titrated up by one tablet (1 matching placebo tablet) per day on a weekly basis until a maximal tolerated dose of at least two tablets (2 placebo tablets) and no more than four tablets (4 placebo tablets) is achieved. Subjects will be maintained at their maximum tolerated dose of between two to four tablets per day (2 to 4 placebo tablets) for the duration of the study. Subjects will be seen at 4 weeks after randomization, at 12 weeks after randomization, and then at study end (week 24 or early termination).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cycloset — Cycloset 1.6 -3.2 mg/day
  Other Names: Bromocriptine Mesylate Quick Release
  Arms: Cycloset (Bromocriptine-QR)
Drug: Placebo — Non-active placebo for cycloset
  Arms: Placebo

SUMMARY:
The main objective is to demonstrate the effects of early dopaminergic activation on the autonomic nervous system in subjects with newly diagnosed vs. established type 2 diabetes. The primary endpoint is the effect of Bromocriptine QR on changes in autonomic function measured by assessing sympathetic and parasympathetic function using conventional measures of autonomic function, including power spectral analysis of heart rate as well as peripheral autonomic function using sudorimetry and laser scanning of peripheral microvascular autonomic control.

DETAILED DESCRIPTION:
This is an interventional, twenty-four week, randomized, double blind, placebo-controlled trial with bromocriptine QR in subjects with newly diagnosed and established type 2 diabetes mellitus (T2DM) to evaluate its effects on the cardiovascular and peripheral autonomic nervous system, as well as on inflammatory markers, the leptin/adiponectin system, hormonal levels of RAS and HPA axis, indices of insulin resistance, and measures of oxidative and nitrosative stress. Forty newly diagnosed diabetes subjects and 40 subjects with established diabetes will be enrolled in the study and each randomized to treatment with bromocriptine-QR or placebo.

Secondary endpoints will demonstrate the effects of dopaminergic activation with Bromocriptine-QR on the regulation of Hypothalamic-Pituitary-Axis (HPA) axis hormones, on the plasma levels of markers of inflammation and oxidative/nitrosative stress in newly diagnosed vs. established type 2 diabetes subjects. The study will evaluate treatment effects on inflammatory markers, the Leptin/Adiponectin system, and hormonal levels of rennin-angiotensin system (RAS), aldosterone and cortisol. Specifically, the following markers of inflammation and oxidative/nitrosative stress: 1) C reactive protein (CRP), 2) interleukin-6, 12, and 10, 3) tumor necrosis factor (TNFalpha), 4) plasminogen activator inhibitor (PAI1), superoxide dismutase (SOD), Thiobarbituric acid reactive substances (TBARS) and Asymmetric dimethylarginine (ADMA) will be evaluated. A co-secondary objective of the study will be to assess the impact of Bromocriptine-QR vs Placebo on measures of insulin resistance and glycemic control (e.g., oral glucose tolerance test (OGTT) glucose and insulin, Matsuda index, Homeostasis Model Assessment-insulin resistance (HOMA-IR), Hemoglobin A1c (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes subjects between the ages of 30 and 80 years of age, inclusive, at Screening
* Hemoglobin A1c (HbA1c) ≤10.0% at screening
* Male or female (female of child bearing age must use definitive contraceptive therapy)
* Type 2 Diabetes Mellitus subjects on a stable anti-diabetes regimen of diet and/or metformin alone therapy or on metformin plus an insulin secretion enhancer (sulfonylureas, dipeptidyl peptidase 4 (DPP4) Inhibitors, Glucagon-like peptide (GLP-1) analogs) therapy for a 60 day period prior to randomization. Subjects with diabetes duration of ≥ 4 years must be using an insulin secretion enhancer (e.g. sulphonylureas (SU), DPP4, GLP-1 analog). Subjects must have a documented C-peptide level (either fasting or random) of >2 ng/ml from the screening visit.

Exclusion Criteria:

* Presence of type 1 diabetes mellitus (defined as C-peptide <1 ng /ml)
* Type 2 diabetes mellitus subjects on insulin.
* Use of prescription sympathomimetics, ergot alkaloid derivatives, or anti-migraine medications, dopamine2 (D2)-like receptor antagonists (e.g. metoclopramide, domperidone) or systemic corticosteroids
* Uncontrolled hypertension (systolic BP >160 or diastolic BP > 100 at screening) or a history of orthostatic hypotension
* History of significant gastroparesis
* Presence of diabetic retinopathy that is more severe than "background" level
* Presence of diabetic nephropathy, or renal impairment defined by blood urea nitrogen (BUN) >40mg/dl and serum creatinine > 1.4 mg/dl if female taking metformin, >1.5 mg/dl. if male taking metformin, and >1.6 mg/dl if not taking metformin
* Presence of clinically significant peripheral or autonomic neuropathy that is clearly of non-diabetic origin
* History of major macrovascular events such as myocardial infarction or cerebrovascular event such as stroke within the past 6 months. Other exclusions include coronary artery bypass graft or coronary angioplasty in the previous 3 months, unstable angina pectoris (chest pain at rest, worsening chest pain, or admission to the emergency room or hospital for chest pain) within the previous 3 months, or seizure disorders.
* Active infection (e.g., human immunodeficiency virus (HIV), hepatitis), or a history of severe infection during the 30 days prior to screening
* Major surgical operation during the 30 days prior to screening
* Cancer, other than non-melanoma skin or non-metastatic prostate cancer, within the past 5 years
* Uncontrolled or untreated hypothyroidism as evidenced by thyroid stimulating hormone (TSH) concentrations >4.8 µU/ml
* Other serious medical conditions which, in the opinion of the investigator, would compromise the subject's participation in the study, including any concurrent illness, other than diabetes mellitus, not controlled by a stable therapeutic regimen, or conditions or abnormalities (e.g., blindness) that might interfere with interpretation of safety or efficacy data, or history of non-compliance
* Clinically significant abnormalities on screening laboratory evaluation, unless approved by the Sponsor
* Abnormalities of liver function defined as any liver enzymes (aspartate aminotransferase (AST), alanine aminotransferase (ALT), serum glutamic-pyruvic transaminase (SGPT), Serum glutamic oxaloacetic transaminase (SGOT) greater than 3 times the upper limit of normal
* History of New York Heart Association (NYHA) Class III-IV congestive heart failure.
* Concurrent participation in another clinical trial with use of an experimental drug or device within 30 days of study entry.
* History of alcohol or substance abuse or dementia
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening. Women who become pregnant will be discontinued from the study.
* Known hypersensitivity to any of the formulation components
* Working rotating, varying or night shifts
* Use of unapproved herbal supplements that may be associated with a risk of cardiovascular events (such as ephedra, yohimbe etc)
* Patients who have started therapy with an erectile dysfunction drug within 2 weeks prior to screening; patients may not begin treatment with an erectile dysfunction drug during the study period; patients currently taking erectile dysfunction drugs should do so only under medical supervision.
* Donation of blood in the previous 30 days. Blood donation is also not allowed during the study or for 30 days after completion of the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virgnia Medical School, Strelitz Diabetes Center, Norfolk, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and thirteen subjects were screened between 05OCT2015 and 29MAR2018 at Eastern Virginia Medical School Endocrine and Metabolic Disorders Outpatient Clinic
Pre-assignment Details: Of the 113 patients screened, 29 screened failed and 84 were enrolled
Groups:
- Cycloset (Bromocriptine-QR): Subjects were randomized in a double blind 1:1 ratio to receive UDT (usual diabetes therapy) plus bromocriptine-QR. Following randomization subjects were titrated to the maximum tolerated dose of the study drug over a four-week period. During these first 4 weeks, the daily dose of the study drug was titrated up by one tablet (0.8 mg bromocriptine-QR) per day on a weekly basis until a maximal tolerated dose of at least two tablets (1.6 mg/day bromocriptine-QR) and no more than four tablets (3.2 mg/per day b-QR) was achieved. Subjects were maintained at their maximum tolerated dose of between two to four tablets per day (1.6 to 3.2 mg bromocriptine-QR per day) for the duration of the study (24 weeks). Subjects were evaluated at 4 weeks after randomization, at 12 weeks after randomization, and then at study end (week 24 or early termination).
  Cycloset: Cycloset 1.6 -3.2 mg/day
- Placebo: Subjects were randomized in a double blind 1:1 ratio to receive UDT (usual diabetes therapy) plus placebo. Following randomization subjects were titrated to the maximum tolerated dose of the study drug over a four-week period. During these first 4 weeks, the daily dose of the study drug was titrated up by one tablet (1 matching placebo tablet) per day on a weekly basis until a maximal tolerated dose of at least two tablets (2 placebo tablets) and no more than four tablets (4 placebo tablets) was achieved. Subjects were maintained at their maximum tolerated dose of between two to four tablets per day (2 to 4 placebo tablets) for the duration of the study. Subjects were evaluated at 4 weeks after randomization, at 12 weeks after randomization, and then at study end (week 24 or early termination).
  Placebo: Non-active placebo for cycloset
Period: Overall Study
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Started | 43 | 41
Completed 4 Weeks | 38 | 39
Completed 12 Weeks | 36 | 37
Completed | 33 | 37
Not Completed | 10 | 4
Not completed — Adverse Event | 10 | 3
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.01 (10.39) | 61.92 (11.55) | 60.43 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 12 | 18 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 22 | 47
  White | 17 | 19 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 43 | 41 | 84
Duration of Diabetes [Median (Inter-Quartile Range); unit: Years] | 8 [3 to 13] | 10 [6 to 15.5] | 8.5 [4.63 to 15]
Height [Mean (Standard Deviation); unit: Inches] | 66.69 (4.08) | 67.19 (3.63) | 66.93 (3.85)
Weight [Mean (Standard Deviation); unit: Pounds] | 214.81 (57.63) | 225.12 (47.57) | 219.84 (52.89)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 33.55 (6.96) | 35.05 (7.87) | 34.28 (7.41)
Percent Body Fat [Mean (Standard Deviation); unit: percentage of body fat] | 39.09 (6.13) | 39.86 (7.55) | 39.45 (6.80)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131.62 (15.22) | 133.93 (16.17) | 132.76 (15.65)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 82.19 (10.65) | 82.07 (9.11) | 82.13 (9.86)
Heart Rate [Mean (Standard Deviation); unit: Beats per minute] | 80.91 (14.65) | 75.29 (10.96) | 78.17 (13.21)

OUTCOME MEASURES:

1. Primary Outcome: Change in E/I Ratio From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: Cardiac Autonomic Reflex Tests (CARTs) based on heart rate variations are the deep breathing test (E/I ratio), the lying to standing test (30:15 ratio) and the Valsalva maneuver (Valsalva ratio). These tests require a continuous recording of heart rate by either a simple electrocardiograph (ECG), subsequently elaborated via a specialist software. It is essential to inspect the ECG trace (on paper or monitor) in order to exclude artifacts or any type of arrhythmias from the calculations.
  Expiration/Inspiration (E/I) ratio: Standardized CART that measures parasympathetic control of the HR. The subject in a supine or sitting position is asked to breathe deeply at six breaths per minute (5 seconds in and 5 seconds out) for one minute. The E/I ratio is obtained by calculating the ratio between the average of the 3 longest RR intervals during expiration and the average of the 3 shortest RR intervals during inspiration.
Time Frame: Baseline to 24 weeks
Population: All participants who completed the study and received 24 weeks of intervention (33 subjects in the bromocriptine QR arm and 37 subjects in the placebo arm)
Measure: Mean (95% Confidence Interval); unit: E/I ratio change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
E/I ratio change | -0.02 [-0.05 to 0.04] | -0.05 [-0.15 to 0.02]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.603, t-test, 2 sided — Between treatment group (bromocriptine-QR vs. placebo) differences in change from baseline to week 24 was analyzed using Independent Samples T-tests. Means are statistically significantly different at the 5% level (P < 0.05) two-sided

2. Primary Outcome: Change in Valsalva Ratio From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: Cardiac Autonomic Reflex Tests (CARTs) based on heart rate variations are the deep breathing test (E/I ratio), the lying to standing test (30:15 ratio) and the Valsalva maneuver (Valsalva ratio). These tests require a continuous recording of heart rate by simple electrocardiograph (ECG), subsequently elaborated via a specialist software. It is essential to inspect the ECG trace (on paper or monitor) in order to exclude artifacts or any type of arrhythmias from the calculations.
  Valsalva maneuver is a forced expiration with an open glottis against resistance. This causes changes in both BP and heart rate. During strain, tachycardia is initially determined by vagal withdrawal and afterwards by sympathetic activation. The Valsalva ratio is calculated as the ratio between the longest RR interval after the expiratory straining and the shortest RR interval during the expiratory straining
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Valsalva ratio change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
Valsalva ratio change | -0.02 [-0.14 to 0.09] | 0.02 [-0.04 to 0.08]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.068, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Change in 30:15 Ratio From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: Lying to Standing (30:15) ratio: HR increases after standing to maintain an appropriate stroke volume, and then decreases. The maximum increase in heart rate generally occurs between the 10th and the 20th beat after standing, whereas heart rate generally returns to lower values between the 25th and the 35th beat. After lying in the supine position for at least 5 minutes, the subject is invited to stand up quickly but remain relaxed for 3 to 5 minutes. The ratio is the longest RR interval measured between the 25th and the 35th beat divided by the shortest RR interval measured between the 10th and the 20th beat after standing up.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: 30:15 ratio change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
30:15 ratio change | -0.03 [-0.06 to 0.001] | -0.02 [-0.04 to 0.006]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.493, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

4. Primary Outcome: Change in SDNN From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: Time domain analysis of Heart Rate Variability includes SDNN and RMSSD measurements. It is acquired by continuous recording of heart rate by simple electrocardiograph (ECG) with the subject in supine or sitting position, resting and breathing at a controlled rate (15 breaths per minute) for 5 minutes. It is essential to inspect the ECG trace in order to exclude artifacts or any type of arrhythmias from the calculations.
  SDNN is the standard deviation of the beat to beat (NN) variability which is a measure of both sympathetic and parasympathetic action on HR.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Milliseconds (ms) change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
Milliseconds (ms) change | -3.97 [-9.20 to 1.26] | -0.80 [-9.14 to 7.54]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.524, t-test, 2 sided — Between treatment group (bromocriptine-QR vs. placebo) differences in change from baseline to week 24 was analyzed using Independent Samples T-tests. Means were statistically significantly different at the 5% level (P < 0.05) two-sided

5. Primary Outcome: Change in RMSSD From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: Time domain analysis of Heart Rate Variability includes SDNN and RMSSD measurements. It is acquired by continuous recording of heart rate by simple electrocardiograph (ECG) with the subject in supine or sitting position, resting and breathing at a controlled rate (15 breaths per minute) for 5 minutes. It is essential to inspect the ECG trace in order to exclude artifacts or any type of arrhythmias from the calculations.
  RMSSD is the root mean square of successive R-R intervals and is a measure primarily of parasympathetic activity on HR.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Milliseconds (ms) change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
Milliseconds (ms) change | -3.16 [-9.08 to 2.76] | -0.57 [-9.43 to 8.29]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.630, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

6. Primary Outcome: Change in Resting Heart Rate From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: The primary outcome is the change from baseline to endpoint (24 weeks) in measures of autonomic function using provocative tests (CARTs), measures of heart rate variability and resting heart rate
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: beats per minute change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
beats per minute change | -0.73 [-3.66 to 2.14] | -2.00 [-4.96 to 0.96]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.537, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

7. Primary Outcome: Change in Feet ESC From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: The coprimary outcome is the change, from baseline to endpoint (24 weeks), of peripheral autonomic function using sudorimetry. Sudoscan measures the sweating capacity of palms and soles and is expressed as electrochemical skin conductance (ESC) of feet and hands. ESC, expressed in micro-Siemens (µS), is the ratio between the current generated and the constant direct voltage stimulus applied to palms and soles between the electrodes. ESC is dependent on the glands' capability to transfer chloride ions and reflects small-C fiber function.
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microSiemmens (µS) change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
microSiemmens (µS) change | -2.40 [-8.59 to 3.79] | -4.57 [-8.32 to -0.82]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.530, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

8. Primary Outcome: Change in Hands ESC From Baseline to Endpoint After 24 Weeks of Intervention With Bromocriptine QR vs Placebo
Description: as for outcome 7
Time Frame: Baseline to 24 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: microSiemmens (µS) change
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
Number analyzed (Participants) | 33 | 37
microSiemmens (µS) change | -1.71 [-5.37 to 1.95] | -9.83 [-14.03 to -5.64]
Statistical Analysis 1: Comparison: Cycloset (Bromocriptine-QR) vs Placebo; Test type: Superiority; p = 0.005, t-test, 2 sided — [p-value comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Cycloset (Bromocriptine-QR) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/41
Serious Adverse Events (participants affected / at risk) | 3/43 | 2/41
Other Adverse Events (participants affected / at risk) | 7/43 | 2/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycloset (Bromocriptine-QR) (N=43) | Placebo (N=41)
Vasovagal Syncope (Nervous system disorders) | 1 (1) | 0 (0) — Vasovagal Syncope secondary to Valsalva maneuver
Acute Metabolic Encephalopathy (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Acute Metabolic Encephalopathy secondary to dehydration with consequent acute kidney failure and rhabdomyolisis
Motor vehicle accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural and Pericardial Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cycloset (Bromocriptine-QR) (N=43) | Placebo (N=41)
Fatigue (General disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT02682901/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/01/NCT02682901/SAP_001.pdf